CLINICAL TRIAL: NCT02377310
Title: A Comparative Study of Resting Coronary Pressure Gradient, Instantaneous Wave-free Ratio and Fractional Flow Reserve in an Unselected Population Referred for Invasive Angiography: The VERIFY 2 Study
Brief Title: Pd/Pa vs iFR™ in an Unselected Population Referred for Invasive Angiography
Acronym: VERIFY2
Status: Completed | Type: Observational
Sponsor: Golden Jubilee National Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 1.0
Record Dates: First submitted 2015-02-26; First posted 2015-03-03 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Coronary Artery Disease; Plaque; Atherosclerosis; Fractional Flow Reserve
MeSH Terms: conditions — Coronary Artery Disease; Plaque, Amyloid; Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All patients: All patients will undergo coronary physiological study with measurement of resting Pd/Pa, iFR™, hyperaemic iFR and FFR.

SUMMARY:
Instantaneous wave-free ratio (iFR™) is a novel non-hyperaemic index of the functional significance of a coronary stenosis. Previous studies have shown variable levels of correlation with the established hyperaemic index FFR. In addition it has been proposed that iFR™ has superior diagnostic accuracy when compared to mean whole cardiac cycle Pd/Pa which can also be used to predict FFR.

We plan to undertake a prospective clinical study in consecutive patients already undergoing FFR assessment in the cardiac catheterisation laboratory to compare the ability of iFR™ and Pd/Pa (both measured using the proprietary Volcano system) to predict FFR. We will explore the level of misclassification of flow limiting disease that results from use of iFR™ and resting Pd/Pa employed using either binary cut-off algorithms or in a hybrid decision making protocol. We plan to analyse 260 vessels over a 18 month period. Hyperaemia will be induced by intravenous adenosine (140 ug/kg/min) administered wherever possible via an antecubital vein. Intra-coronary nitrates will also be given in line with the standard care procedure for FFR measurement. Final clinical decisions following coronary physiology will be based on steady state FFR.

DETAILED DESCRIPTION:
Title:

A comparative study of resting Pd/Pa, instantaneous wave-free ratio and fractional flow reserve in an unselected population referred for invasive angiography.

Instantaneous wave-free ratio (iFR™) is a novel non-hyperaemic index for assessing the functional significance of a coronary stenosis without coronary vasodilatation. In previous studies it has been compared to the hyperaemic index FFR with variable results. As a guide to determining the need for revascularisation it has been employed using a dichotomous cut-off without FFR or within a hybrid strategy in which lesions with intermediate iFR™ values are further interrogated using FFR.

The comparative diagnostic utility of iFR™ vs resting pressure (Pd/Pa) in reference to FFR is uncertain. We plan to undertake a prospective clinical study in consecutive patients undergoing clinically-indicated FFR assessment in the cardiac catheterisation laboratory with 30-80% diameter stenosis on quantitative coronary angiography (QCA). We will will use a proprietary (Volcano) pressure wire system and iFR ™ algorithm in order to calculate iFR™ and Pd/Pa in both resting and hyperemic conditions as well as FFR.

The sample size is 260 vessels and the enrolment period is 18 months. Hyperaemia will be induced by intravenous adenosine (140 ug/kg/min) administered wherever possible via an antecubital vein. Intra-coronary nitrates will also be given in line with the standard care procedure for FFR measurement.

Design:

In this prospective single centre cohort study all consecutive patients undergoing FFR are eligible for inclusion.

Active Hypothesis: (1) In comparison to an FFR for all strategy, revascularisation decisions made using binary cut-off values of iFR™ or resting Pd/Pa will result in similar levels of disagreement.

Active Hypothesis: (2) In comparison to an FFR for all strategy, revascularisation decisions using hybrid strategies incorporating iFR™ or resting Pd/Pa and FFR will result in similar levels of disagreement.

Active Hypothesis (3): Compared to iFR™ measured under resting conditions, hyperaemic iFR™ has a stronger correlation with FFR. Should this be the case, then the diagnostic efficiency of iFR™ can be interpreted as being improved with pharmacological vasodilatation. The null hypothesis is that there is no difference in diagnostic efficiency between iFR™ and hyperaemic iFR compared to FFR.

The clinical decisions in the catheter laboratory will align with routine care and be informed by all available clinical data and the FFR results.

This study is being conducted independently in the National Health Service without industry support or involvement.

Sample size: 260 vessels.

Statistical Analysis: Independent analysis of the completed dataset will be performed by Dr John McClure a biostatistician and lecturer in the Institute of Cardiovascular and Medical Sciences in Glasgow.

Methods: We will measure resting indices Pd/Pa and iFR™. Following this we will then measure hyperaemic readings including FFR and hyperaemic iFR™ (HiFR) sequentially using peripherally administered adenosine. Upon completion of enrollment we will produce summary statistics describing demographics and procedural data for the study cases. We will then calculate the discriminatory power of iFR™ using both the pre-specified binary cut-off values of 0.90 for iFR™ and 0.92 for resting Pd/Pa and the adenosine zones for iFR of 0.86-0.93 and resting Pd/Pa of 0.87-0.94. We will also analyse the correlation of HiFR with FFR

ELIGIBILITY:
Inclusion Criteria:

All patients ≥18 years of age, already undergoing pressure wire assessment and able to consent

Exclusion Criteria:

Inability to receive adenosine

Extremely tortuous vessels

Highly calcified lesions unsuitable for pressure wire assessment

coronary artery occlusion

acute MI within 3 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients undergoing FFR assessment for standard clinical indications.
Sampling Method: Non-Probability Sample
Enrollment: 197 (Actual)
Dates: Start 2013-09; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
To determine the diagnostic accuracy of instantaneous wave-free ratio (binary cut-off value 0.90) versus resting Pd/Pa (binary cut-off value 0.92) in reference to FFR. | 30 days
  Resting Pd/Pa will be compared to iFR™ in reference to FFR.

SECONDARY OUTCOMES:
To determine the diagnostic accuracy of hybrid iFR™/FFR versus hybrid resting Pd/Pa/FFR in reference to FFR | 30 days
  Adenosine zone for iFR is 0.86-0.93, Adenosine zone for resting Pd/Pa is 0.87-0.94.
To compare steady state FFR to minimum FFR | 30 days
  FFR recorded by the operator as the minimum value will be compared with the steady state value and the impact on vessel classification will be assessed
To investigate the influence of hyperemia on iFR™. | 30 days
  iFR™ will be reassessed after administration of adenosine to evaluate whether this increases agreement with FFR.
To assess the rate of revascularization per (1) artery and (2) per patient, associated with iFR™-guided management vs. FFR-guided management. | 30 days
  An analysis of the total number of vessels and patients that would potentially undergo revascularisation will be used to compare iFR™ versus FFR guided managment.
To assess serious adverse events in patients receiving intravenous adenosine | 30 days
  Patients will be monitored during coronary physiology studies to assess the safety of intravenous adenosine infusion with assessment of side effects leading to early termination of the infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Keith G Oldroyd, M.D., Study Director — Golden Jubilee National Hospital
Locations (1):
- Golden Jubilee National Hospital, Glasgow, Dunbartonshire, United Kingdom

REFERENCES:
- [Background] Bossuyt PM, Reitsma JB, Bruns DE, Gatsonis CA, Glasziou PP, Irwig LM, Lijmer JG, Moher D, Rennie D, de Vet HC; Standards for Reporting of Diagnostic Accuracy. Towards complete and accurate reporting of studies of diagnostic accuracy: the STARD initiative. Clin Radiol. 2003 Aug;58(8):575-80. doi: 10.1016/s0009-9260(03)00258-7. PMID 12887949
- [Derived] Van't Veer M, Pijls NHJ, Hennigan B, Watkins S, Ali ZA, De Bruyne B, Zimmermann FM, van Nunen LX, Barbato E, Berry C, Oldroyd KG. Comparison of Different Diastolic Resting Indexes to iFR: Are They All Equal? J Am Coll Cardiol. 2017 Dec 26;70(25):3088-3096. doi: 10.1016/j.jacc.2017.10.066. PMID 29268922
- [Derived] Hennigan B, Oldroyd KG, Berry C, Johnson N, McClure J, McCartney P, McEntegart MB, Eteiba H, Petrie MC, Rocchiccioli P, Good R, Lindsay MM, Hood S, Watkins S. Discordance Between Resting and Hyperemic Indices of Coronary Stenosis Severity: The VERIFY 2 Study (A Comparative Study of Resting Coronary Pressure Gradient, Instantaneous Wave-Free Ratio and Fractional Flow Reserve in an Unselected Population Referred for Invasive Angiography). Circ Cardiovasc Interv. 2016 Nov;9(11):e004016. doi: 10.1161/CIRCINTERVENTIONS.116.004016. PMID 27834663